CLINICAL TRIAL: NCT07127393
Title: Sensory Evaluation of Foods Formulated With Seaweeds and Their Effect on Satiety and Food Intake
Brief Title: Adding Chondrus Crispus Seaweeds to a Meal: Effect on Sensory Perception, Physical Comfort, Satiety and Food Intake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: Acadian Seaplants (Unknown)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-001
Record Dates: First submitted 2025-08-06; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Satiety and Food Intake; Sensory Evaluation; Physical Comfort
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal with seaweed (Experimental): Omelette with added Chondrus crispus seaweeds
  Interventions: Other: Food
- Meal without seaweed (Experimental): Omelette
  Interventions: Other: Food
- Water Control (Experimental): Potable water
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Meal with seaweed

SUMMARY:
The study investigates the sensory characteristics, consumer perception and the effect on satiety and food intake of the meal with added Chondrus crispus seaweed produced by Acadian Seaplants in Atlantic Canada.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adult males

Exclusion Criteria:

* Having any diseases
* Smoking, consuming cannabis
* Skipping breakfast regularly
* Disordered eating patterns
* Taking certain medications that may affect the central and peripheral mechanisms of food intake regulation, cognitive performance and sedative medications
* Food allergies and aversion towards seaweeds

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Appetite | 0-120 minutes
  The average subjective appetite is a result of the desire to eat, hunger, prospective food consumption, and fullness.
Food Intake | 120 minutes
  Ad libitum food intake is being measured with crustless pizza until the participants feel comfortably full.

SECONDARY OUTCOMES:
Physical Comfort | 0-120 minutes
  The subjective feelings of gastrointestinal discomfort, wellness, perceived energy, and fatigue levels.
Mastication | 5 minutes
  The number of chewing cycles per bite.
Taste and other sensory characteristics | 0, 120 minutes
  The hedonic and intensity perceptions, including pleasantness, taste, texture, chewing, and other sensory characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Appetite Lab, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No